CLINICAL TRIAL: NCT01658423
Title: EFFECT OF MATURITY ON SPRINT AND JUMP PERFORMANCES IN ADOLESCENT BOYS.
Brief Title: Maturity and Motor Fitness
Acronym: MMF
Status: Completed | Type: Observational
Sponsor: National Institute of Fitness and Sports in Kanoya (Other)
Collaborators: Junior high school (Unknown)
Responsible Party: Principal Investigator, Yohei Takai, Assisstant Professor, National Institute of Fitness and Sports in Kanoya
Other Study IDs: NIFS-002
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Physical Fitness
Keywords: pubic hair; sprint velocity; vertical jump height; body composition; maximal voluntary torque

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Junior high school student: All subjects participated in measurements of body composition, muscle strength and motor fitness

SUMMARY:
The current study examined the effect of maturity on the sprint and jump performances in a single year age group of 13 year old boys.

DETAILED DESCRIPTION:
The investigators examined the issue in adolescent boys (n = 107) aged from 13.0 to 13.9 years. The maturity status was assessed using a self-assessment of stage of pubic hair based on the criteria of Tanner. Body composition and maximal voluntary knee extension torque (KET) were determined using a bioelectrical impedance analyzer and a static myometer, respectively. Sprint velocity was measured by a non-motorized treadmill. Jump height was calculated from the following equation; g × (flight time)2 × 8 × 10-1. The flight time during jumping was measured by a matswitch system.

ELIGIBILITY:
Inclusion Criteria:

* adolescents

Exclusion Criteria:

* subjects had some diseases and disorders

Ages: 156 Months to 167 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Junior high school students
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2011-03; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 day
  Bioelectrical impedence - percent body fat

SECONDARY OUTCOMES:
Muscle strength | 1 day
  myometer- knee extension strength

CONTACTS AND LOCATIONS:
Locations (1):
- Chosa junior high school, Kokubu-matsuki, Kagoshima-ken, Japan

REFERENCES:
- [Background] Armstrong N, Welsman JR, Chia MY. Short term power output in relation to growth and maturation. Br J Sports Med. 2001 Apr;35(2):118-24. doi: 10.1136/bjsm.35.2.118. PMID 11273974